CLINICAL TRIAL: NCT01708148
Title: Oral Administration of Four Lactobacillus Species Preparation to Improve the Quality of the Neovaginal Flora in Male to Female Transsexual Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: University of Natural Resources and Life Sciences, Vienna, Austria (Other)
Responsible Party: Principal Investigator, Associate Prof. Ljubomir Petricevic MD, Ass. Prof MD, Medical University of Vienna
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: MUW EK982/2010
Record Dates: First submitted 2012-10-11; First posted 2012-10-16 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Reduction or Absence of Lactobacilli in Neovaginal Flora
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactobacilli (Active Comparator): 30 Participants with verum
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): 30 Participants
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — lyophilised L. rhamnosus, L. jensenii, L. crispatus, L. gasseri and sodium alginate
  Arms: Lactobacilli
Other: Placebo — control group would receive a oral lactose placebo
  Arms: Placebo

SUMMARY:
The aim of this study is the improvement of the penile linked neovaginal flora in male-to-female transsexuals after application of oral probiotics.

ELIGIBILITY:
Inclusion Criteria:

Participants underwent the sex reassignment surgery (SRS) with the technique of the inverted penile skin flap longer than 1 year.

All transsexual women treated according to the Standards of Care of the World Professional Association of Transgender Health (WPATH).

Exclusion Criteria:

* clinical signs of vaginal or urinary tract infection,
* abnormal neovaginal discharge,
* neoplasia,
* bleeding,
* diarrhoea,
* constipation,
* rectal pathologies including hemorrhoids,
* antibiotic therapy in the previous 4 weeks

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
change in Nugent score between baseline and end of treatment (improvement or no improvement). | day 0 day 7 of oral probiotic application
  Using Nugent scoring system, from each participant first swab from neovagina and rectum will be taken before start of oral probiotic use.(baseline information) Second swab from neovagina and rectum will be taken on the day following the last administration.(information about change in Nugent)

SECONDARY OUTCOMES:
Isolation of specific Lactobacilli from neovaginal microbiologic cultures after oral administration of probiotic | Day 7 of oral probiotic application
  From each participant, the swab from neovagina and rectum for microbiologic cultures will be taken on the day following the last administration. Isolation of oral applied probiotic strains.

OTHER OUTCOMES:
Nugent Score | day 0 day 7 of oral probiotic application

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gyecology, AKH, Vienna, Vienna, Austria